CLINICAL TRIAL: NCT06331975
Title: Radiomics and Radiogenomics of Non-small Cell Lung Cancer: Relationships of Radiomic Signature With Gene Driver Mutations and Implications for Emerging Therapies
Brief Title: Radiomics and Radiogenomics of Non-small Cell Lung Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: European Institute of Oncology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IEO 0836
Record Dates: First submitted 2024-03-18; First posted 2024-03-26 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Radiomic signature (Other): Assessment of radiomic signature and tumor genetic profile at baseline
  Interventions: Diagnostic Test: Radiomic signature

INTERVENTIONS:
Diagnostic Test: Radiomic signature — Assessment of radiomic signature and tumor genetic profile in patients with Non Small Cell Lung Cancer (NSCLC)

SUMMARY:
In this study, the radiomic characteristics and a broad range of genetic aberrations in lung adenocarcinomas will be evaluated. Investigators will assess changes in the radiomic and genetic profiles during targeted therapies in a subset of patients harboring treatable mutations. Patients undergoing targeted therapies will also be evaluated for variations in genomic profile and radiomic signature during follow-up

DETAILED DESCRIPTION:
Non-small cell lung cancers (NSCLC) are the first cause of cancer-related deaths.

Recent guidelines suggest the key role of a wide molecular profile because knowledge of the tumor genotype can enable patients with NSCLC to be treated with targeted therapies.

In this study, a first group of patients with lung adenocarcinoma (study group), tested for the presence of genetic alterations in EGFR, ALK, and KRAS, and with available Computer Tomography (CT) scans, will be evaluated to create a radiomic signature and assess its association with mutational status and prognosis.

Then, a second group of patients (validation group) will be enrolled to validate the radiomic signature and the status of the genetic alterations and their association with prognosis. Radiomic signature and liquid biopsies will be evaluated in patients positive for genetic alterations at each follow-up step to verify their association with prognosis and response to targeted therapies.

ELIGIBILITY:
Inclusion Criteria:

* patients with diagnosis of NSCLC
* patients candidates for mutational status assessment

Exclusion Criteria:

- patients with age <18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2018-06-12 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-09-14 (Actual)

PRIMARY OUTCOMES:
Evaluation of the association between the status of Epidermal Growth Factor Receptor (EGFR), Anaplastic Lymphoma Kinase (ALK), Kirsten Rat Sarcoma Virus (KRAS) and nodal status | 1 month
  The status of EGFR, ALK, KRAS will be validated for its association with nodal status at surgery
Evaluation of the association between the status of EGFR, ALK, KRAS and overall survival (OS) | 5 years
  Number of patiens with EGFR, ALK, KRAS mutations alive at five years
Evaluation of the association between the status of EGFR, ALK, KRAS and disease free survival (DFS) | 5 years
  Number of patiens with EGFR, ALK, KRAS mutations with an oncological event (local or distant) during follow up

CONTACTS AND LOCATIONS:
Overall Officials: Francesca Botta, Principal Investigator — European Institute of Oncology
Locations (1):
- European Institute of Oncology, Milan, Italy